CLINICAL TRIAL: NCT02395211
Title: Effects of Proprioceptive Stimulation Under Visual Feedback in Patient With CRPS: An Exploratory Study
Brief Title: Effects of Proprioceptive Stimulation Under Visual Feedback in Patient With CRPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Studio_CRPS_gloreha
Record Dates: First submitted 2015-03-16; First posted 2015-03-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Physiotherapy (Active Comparator)
  Interventions: Behavioral: Usual Physiotherapy
- Gloreha device (Experimental)
  Interventions: Device: Gloreha device

INTERVENTIONS:
Behavioral: Usual Physiotherapy — Usual physiotherapy consist of active or passive mobilization, extensor digiti and carpi functional electric stimulation, occupational therapy and taping.
  The intervention will last 30 minute a day x 4 weeks
  Arms: Usual Physiotherapy
Device: Gloreha device — Proprioceptive stimulation under visual feedback are provided by the Gloreha device. The intervention will last 30 minute a day x 4 weeks
  Arms: Gloreha device

SUMMARY:
The aim of this study is to evaluate feasibility of a proprioceptive stimulation under visual feedback treatment protocol (using Gloreha® device) compared to usual physiotherapy treatment in sub-acute stroke patient with Complex regional pain syndrome.

DETAILED DESCRIPTION:
The aim of this study is to evaluate feasibility of a a proprioceptive stimulation under visual feedback treatment protocol (using Gloreha® device) compared to usual physiotherapy treatment in sub-acute stroke patient with Complex regional pain syndrome.

Treatments effect will be evaluated on pain perception, upper extremity functionality and change in pain pressure treshold.

Usual physiotherapy consist of active or passive mobilization, extensor digiti and carpi functional electric stimulation, occupational therapy and taping.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years and < 85 years
* diagnosis of stroke < 6 months prior to study enrollment
* diagnosis of Complex regional pain syndrome according to Budapest Criteria

Exclusion Criteria:

* neurological or psychiatric pathology
* severe cardio-pulmonary, renal, hepatic diseases
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Change measures (weeks: 0,4,16, 28)

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | Change measures (weeks: 0,4,16, 28)
McGill Pain Questionnaire | Change measures (weeks: 0,4,16, 28)
  The MPQ is a self-report measure of pain studied with a number of diagnoses. The MPQ assesses both the quality and intensity of subjective pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain.
Erasmus MC modification to the (revised) Nottingham Sensory Assessment - Italian version | Change measures (weeks: 0,4,16, 28)
Fugl-Meyer Upper Extremity | Change measures (weeks: 0,4,16, 28)
  Measure of upper extremity motor impairment. The upper extremity score ranges from 0-66
Pressure Pain Threshold | Change measures (weeks: 0,4,16, 28)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Ferrara, Italy